CLINICAL TRIAL: NCT04228367
Title: JuggerStitch™ for Meniscal Repair Post Market Clinical Follow-up Study
Brief Title: JuggerStitch Post Market Clinical Follow-up Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CMG2017-14SM
Record Dates: First submitted 2020-01-10; First posted 2020-01-14 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Meniscus Tear, Tibial; Meniscus Lesion
MeSH Terms: conditions — Tibial Meniscus Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Meniscal repair (Experimental): Patients in need of meniscal repair
  Interventions: Device: JuggerStitch Meniscal Repair Device

INTERVENTIONS:
Device: JuggerStitch Meniscal Repair Device — Treatment of torn meniscus with JuggerStitch.

SUMMARY:
This study is a post-market follow-up study. The data collected from this study will serve the purpose of confirming the safety and performance of the JuggerStitch Device used for meniscal repair according to the product labelling (Instruction For Use).

DETAILED DESCRIPTION:
This study is a post-market follow-up study to fulfil the post-market surveillance obligations according to Medical Device Directive and MEDDEV 2.12/2 and the Medical Devices Regulation (MDR 2017/745). The data collected from this study will serve the purpose of confirming the safety and performance of the JuggerStitch Device used for meniscal repair according to the product labelling (IFU).

The objectives of the study are to calculate the overall clinical success rate and the performance, and confirm the safety of the JuggerStitch Meniscal Repair Device. The primary endpoint of this study is defined by the absence of reoperation due to meniscal tear. This will be measured against the success criteria of the absence of reoperation in 90.2% of the cases at one year.

ELIGIBILITY:
Inclusion Criteria:

* Subject qualifies for meniscal repair based on the physical exam and medical history and meets the approved indications for use of the study product;
* Older than 18 years and skeletally mature;
* Willing and able to comply with the study procedures;
* Subject is capable of understanding the doctor's explanations, following his instructions and is able to participate in the follow-up program;
* Subject is able to read and understand the informed consent form (ICF) and has voluntarily provided written informed consent.

Exclusion Criteria:

* Meniscal tears in the avascular zone of meniscus;
* Meniscal tears not suitable for repair because of the degree of damage(marked irregularity and complex tearing) to the meniscus body including degenerative, radial, horizontal cleavage and flap tears;
* Presence of active infection;
* If female, subject is pregnant;
* Subject is vulnerable (prisoner, mentally incompetent or unable to understand what participation to the study entails, a known alcohol or drug abuser, anticipated to be non-compliant);
* The subject is unwilling or unable to give consent or to comply with the follow-up program;
* Subject meets any contraindications of the appropriate Instruction for Use.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2020-09-25 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Clinical Success | 1 year
  The absence of reoperation due to meniscal tear. This will be measured against the success criteria of the absence of reoperation in 90.2% of the cases at one year.

SECONDARY OUTCOMES:
Monitoring of Adverse Events to confirm safety of the meniscal repair device | 1 year
  The safety of the system will be assessed by monitoring the frequency and incidence of adverse events

OTHER OUTCOMES:
Lysholm Knee Scoring Scale | Pre-operatively, 6 weeks, 6 months and 1 year post-surgery
  The scale is used to evaluate the outcomes of meniscus surgery. It consists of items that measure: pain, instability, locking, swelling, limp, stair climbing, squatting, and need for support. Lowest and highest scores are 0 and 100 (better), respectively.
Tegner Activity Level Scale | Pre-operatively, 6 weeks, 6 months and 1 year post-surgery
  The Tegner Activity Level Scale aims to provide a standardized method of grading work and sporting activities and complements Lysholm Knee Scoring Scale. The Scale is based on 10 levels with Level 10 being "Competitive Sports" and Level 0 being "Sick Leave".
International Knee Documentation Committee Subjective Knee Evaluation Form (IKDC) | Pre-operatively, 6 weeks, 6 months and 1 year post-surgery
  The IKDC is used to measure symptoms, function, and sports activity for people with meniscal injuries. Lowest and highest (better) scores are 0 and 100, respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Nesma Bayrich, DDS, Study Chair — Zimmer Biomet; Kim Blick, Study Chair — Zimmer Biomet
Locations (6):
- United States (2):
  - OrthoCarolina, Charlotte, North Carolina
  - OrthoVirginia, Inc., Richmond, Virginia
- Ramsay General de Sante - Hôpital Privé Jean Mermoz - Centre Orthopédique Santy, Lyon, France
- Medizinische Fakultät der Otto-von-Guericke-Universität Magdeburg, Magdeburg, Germany
- Japan (2):
  - Ichihara Hospital, Tsukuba, Ibaraki
  - Tokyo Medical and Dental University Hospital of Medicine, Tokyo

IPD SHARING:
Plan to Share IPD: No